CLINICAL TRIAL: NCT02801253
Title: Prospective Cohort of Patients With Prosthetic Joint Infection
Brief Title: Cohort of Prosthetic Joint Infections
Acronym: COPINS
Status: Recruiting | Type: Observational
Sponsor: Groupe Hospitalier Diaconesses Croix Saint-Simon (Other)
Responsible Party: Principal Investigator, Dr Valerie ZELLER, infectious diseases specialist, Groupe Hospitalier Diaconesses Croix Saint-Simon
Other Study IDs: ID RCB: 2014-A01100-47
Record Dates: First submitted 2016-05-27; First posted 2016-06-15 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Management of prosthetic joint infections (PJI) is a challenging task. These infections include different clinical and microbiological settings calling upon various treatment strategies according to infection type (acute or chronic), bone quality, the involved micro-organism and the patient's general condition and willing.

Treatment of PJI combines surgery and prolonged antibiotic therapy. In some patients with a high operative risk prolonged suppressive antibiotic therapy can be used.

Lack of large prospective studies motivated the conception of this cohort with a long term follow up, regardless to PJI management procedures.

DETAILED DESCRIPTION:
Large prospective cohort study in a French referral center for bone and joint infections.

Population

* all patients who consented to participate in the study with PJI treated with:
* debridement-synovectomy for acute infection
* with one-stage, two-stage exchange arthroplasty for chronic infection
* other procedures (complete removal of the prosthesis) and antibiotic therapy
* patients (non-operated or operated) receiving prolonged suppressive antibiotic therapy

Outcome:

* Follow-up at least 2 years
* Events monitored: reinfection including relapse and new infection, joint revision for mechanical failure, PJI related or non-related death Study duration: 10 years. Recruitment period: 4 years. Maximal duration of data collection: 6 years. Investigator center: monocenter study. Mean patient inclusion per year: 100 patients per year.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 18 years old with hip, knee and or shoulder joint prosthesis who consented to participate in the study with:
* According to musculoskeletal infection society definition: PJI is present when one of the major criteria exists or four out of six minor criteria.

Major Criteria:

* Two positive periprosthetic cultures with phenotypically identical organisms, OR
* A sinus tract communicating with the joint, OR

Minor Criteria:

* Elevated serum C-reactive protein (CRP) AND erythrocyte sedimentation rate (ESR)
* Elevated synovial fluid white blood cell (WBC)
* Elevated synovial fluid polymorphonuclear neutrophil percentage (PMN%)
* The presence of pus in the joint without known cause
* Positive histological analysis of periprosthetic tissue
* A single positive culture

Or a PJI which meets the following three criteria:

* Medical story suggesting prosthetic joint infection.
* The presence of pain either with or without swelling for more than 3 months unrelated to a mechanical cause.
* Germ identification in a single sample of fluid aspiration or tissue culture.

  * Or microbial growth in prosthesis sonication fluid culture greater than 50CFU/ml.

Exclusion Criteria:

* Patient who does not meet eligibility criteria.
* Patient lawfully deprived of his liberty.
* Patient not insured under social security scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients managed in the investigators referral center of bone and joint infection, who meet protocol selection criteria will be included in the study. The investigators expect to recruit 400 patients.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2015-09-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with hip and knee prosthetic joint reinfection (relapse and new infection) and multi-variable analysis of reinfection risk factors | 2 years

SECONDARY OUTCOMES:
Assessment of joint function at one, two, four and 6 years after prosthesis revision with one or two stage exchange arthroplasty. | 1, 2, 4, 6 years
Assessment of mechanical failure rate six years after prosthesis revision with one or two stage exchange arthroplasty | 6 years
Assessment of treatment failure rate in patients with hip and knee PJI 2 years after prolonged suppressive antibiotic therapy in non-operated patients. | 2 years
Assessment of reinfection rate of shoulder PJI two years after prosthesis revision with one or two stage exchange arthroplasty. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: VALERIE ZELLER, Doctorate, Principal Investigator — Groupe Hospitalier Diaconesses Croix Saint-Simon
Locations (1):
- Groupe Hospitalier Diaconesses Croix Saint Simon, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No